CLINICAL TRIAL: NCT01755884
Title: Oral Desensitization to Wheat in Children Over 6 Years of Age With Wheat Allergy
Brief Title: Oral Desensitization to Wheat in School Aged Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: University of Oulu (Other); Oulu University Hospital (Other); Tampere University Hospital (Other); Kuopio University Hospital (Other)
Responsible Party: Principal Investigator, Mika Juhani Mäkelä, MD, PhD, Chief Physician, Helsinki University Central Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ODEW
Record Dates: First submitted 2012-12-19; First posted 2012-12-24 (Estimated); Last update posted 2015-03-20 (Estimated); Status verified 2015-03

CONDITIONS: Wheat Allergy
Keywords: Wheat allergy; Immunotherapy; Desensitization; Food allergy; T cells
MeSH Terms: conditions — Wheat Hypersensitivity; Food Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Wheat oral immunotherapy (Experimental): Well-cooked wheat spaghetti is given daily to the patients starting from a minimal dosage (0,0003 g of wheat protein) and increasing the dosing in every 1-2 weeks until a dosage corresponding the size of one meal.
  Interventions: Dietary Supplement: Wheat oral immunotherapy

INTERVENTIONS:
Dietary Supplement: Wheat oral immunotherapy — Cooked spaghetti

SUMMARY:
The aim of the study is to induce tolerance to wheat in wheat allergic children via oral desensitization therapy. The hypothesis is that oral administration of wheat with increasing dosing will increase the individual threshold for allergic reactivity to wheat protein (i.e. desensitization) and even result in no reactivity (i.e. full tolerance). Along with this, the risk for severe allergic reaction to wheat protein is minimized and the diet of patients can partly or completely be normalized. In addition to clinical measures, the immunological mechanisms of desensitization therapy are studied in detail at cellular and molecular level.

DETAILED DESCRIPTION:
This is a prospective multicenter study investigating the efficacy, safety and immunological mechanisms of oral wheat desensitization therapy in school-aged (6-16 yrs of age) wheat allergic children. Wheat allergic children with avoidance diet, immediate reaction in a recent (less than 4 months) food challenge test for wheat and elevated serum wheat-specific IgE levels are recruited to the study. Patients having uncontrolled asthma, other lung disease, cardiovascular disease or other significant systemic disease and patients having poor compliance are excluded. Well-cooked wheat spaghetti is given daily to the patients starting from a minimal dosage (0,0003 g of wheat protein) and increasing the dosing in every 1-2 weeks until a dosage corresponding the size of one meal. The initial dosage is given and certain defined dosage step-ups are carried out in the hospital outpatient clinic. The patient and parents are prepared for the emergency treatment of severe allergic reaction and carry adequate medication with them. The daily use of spaghetti continues with the received maintenance dosage for additional 3 months, until the clinical evaluation of the patient. Thereafter, the patients are allowed to use also other wheat products. Peripheral venous blood samples are taken before therapy and at 3 months and 1 year follow-up visits after reaching the maintenance dosage. The characteristics and function of isolated peripheral blood mononuclear cells (PBMC) will be specifically tested using flow cytometric methods. The expression levels of cell-specific mRNAs (messenger ribonucleic acid) and cytokines are measured with qRT-PCR (quantitative reverse transcriptase real-time polymerase chain reaction)and flow cytometry based methods. In addition, specific IgE (immunoglobulin E) levels are measured and serum samples are frozen for further testing. Two separate control groups are also recruited. The first group includes patients with previous food-challenge proven IgE-mediated wheat allergy with spontaneous recovery and the current free use of wheat protein in their diet. The second group includes children (6-16 yrs of age) who come to hospital for a minor surgical operation (e.g. minor trauma, circumcision, patellar luxation etc.). Children with asthma, allergy, atopic eczema, any other chronic disease or recent infection (less than 2 weeks ago) are excluded from this group. Peripheral venous blood samples are taken from all control children. The characteristics and function of isolated PBMCs, the expression levels of cell-specific mRNAs and cytokines and specific IgE levels are measured.

ELIGIBILITY:
Inclusion Criteria:

* Elevated serum wheat specific IgE
* Immediate reaction in open oral wheat challenge test
* Diet free from wheat, rye, and barley

Exclusion Criteria:

* Uncontrolled asthma
* Other lung disease
* Cardiovascular disease or other significant systemic disease
* Patients having poor compliance

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2009-08; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Efficacy of oral wheat desensitization | 8 months
  Change in the tolerance to wheat and the amount of daily use of wheat in 3 months after the 5 months oral desensitization therapy.

SECONDARY OUTCOMES:
Efficacy of oral wheat desensitization at 17 months | 17 months
  Change in the tolerance to wheat and the amount of daily use of wheat in 1 year after the 5 months oral desensitization therapy.
Safety of oral wheat desensitization therapy at 8 months | 8 months
  Number of participants with adverse events as a measure of tolerability and safety at 3 months after the 5 months desensitization therapy
Safety of oral wheat desensitization therapy at 17 months | 17 months
  Number of participants with adverse events as a measure of tolerability and safety at 1 year after the 5 months desensitization therapy
Effect of the treatment on the characteristics and function of immune cells | 17 months
  Flow cytometric characterization of the change in the proportions of various T cell subtypes and in the function of these cells in in vitro proliferation and suppression tests between the samples taken before the treatment and 3 and 12 months after the treatment.
Effect of the treatment on the cell specific mRNA expression | 17 months
  qRT-PCR measurement of the change in the expression level of T cell subtype specific mRNA levels between the samples taken before the treatment and 3 and 12 months after the treatment.
Effect of the treatment on the cytokine profile | 17 months
  Flow cytometric measurement of the change in the levels of T cell subtype specific cytokine levels between the samples taken before the treatment and 3 and 12 months after the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Mika J Mäkelä, MD, PhD, Principal Investigator — Helsinki University Central Hospital
Locations (4):
- Finland (4):
  - Helsinki University Central Hospital, Helsinki, Helsinki
  - Kuopio University Hospital, Kuopio, Kuopio
  - University of Oulu, Oulu, Oulu
  - Tampere University Hospital, Tampere, Pirkanmaa